CLINICAL TRIAL: NCT03703830
Title: Effects of Cerebellar Transcranial Current Stimulation Associated With Locomotor Training on Functional Mobility of Subjects With Cerebellar Ataxia
Brief Title: tDCS Associated With Locomotor Training on Functional Mobility of Cerebellar Ataxia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Clinical Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cerebellarataxia_ctDCS_LT
Record Dates: First submitted 2018-10-05; First posted 2018-10-12 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Ataxia, Cerebellar
Keywords: Cerebellum; Transcranial direct current stimulation; Gait ataxia
MeSH Terms: conditions — Cerebellar Ataxia; Gait Ataxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental I (Experimental): Cerebellar transcranial current stimulation associated with locomotor training
  Interventions: Device: Cerebellar transcranial direct current stimulation; Other: Treadmill locomotor training
- Sham comparator I (Sham Comparator): Cerebellar transcranial current stimulation sham associated with locomotor training
  Interventions: Other: Treadmill locomotor training; Device: Sham Cerebellar transcranial direct current stimulation
- Experimental II (Experimental): Cerebello-spinal direct current stimulation associated with locomotor training
  Interventions: Other: Treadmill locomotor training; Device: Cerebello-spinal direct current stimulation
- Sham comparator II (Sham Comparator): Cerebello-spinal direct current stimulation sham associated with locomotor training
  Interventions: Other: Treadmill locomotor training; Device: Sham cerebello-spinal direct current stimulation

INTERVENTIONS:
Device: Cerebellar transcranial direct current stimulation — Cerebellar transcranial direct current stimulation (ctDCS) will be applied during 25 minutes at 2 mA of intensity. Anodal electrode will be positioned 1 cm below inion and cathodal electrode at right deltoid muscle.
  Arms: Experimental I
Other: Treadmill locomotor training — The Treadmill Locomotor Training (TLT) will be performed through speed and step length progression protocol for 25 minutes and combined to ctDCS
Device: Sham Cerebellar transcranial direct current stimulation — Sham Cerebellar transcranial direct current stimulation (ctDCS sham) will be applied during 30 seconds at 2 mA of intensity. Anodal electrode will be positioned 1 cm below inion and cathodal electrode at right deltoid muscle. However, subjects will keep the placement of electrodes for 25 minutes to ensure stimulation's masking.
  Arms: Sham comparator I
Device: Cerebello-spinal direct current stimulation — Cerebello-spinal transcranial direct current stimulation (csDCS) will be applied during 25 minutes at 2 mA of intensity. The anode was placed on the scalp over the cerebellum area (1 cm below the inion) and the cathode over the spinal lumbar enlargement (2 cm under T11)
  Arms: Experimental II
Device: Sham cerebello-spinal direct current stimulation — Sham cerebello-spinal direct current stimulation (csDCS sham) will be applied during 30 seconds at 2 mA of intensity. The anode was placed on the scalp over the cerebellum area (1 cm below the inion) and the cathode over the spinal lumbar enlargement (2 cm under T11). However, subjects will keep the placement of electrodes for 25 minutes to ensure stimulation's masking.
  Arms: Sham comparator II

SUMMARY:
Cerebellar ataxia is a neurologic symptom caused by a damage or a dysfunction in cerebellum and results in loss of coordination, balance and postural control. This impairment could result in a reduction of walking speed, short and irregular steps and difficulty in coordinating between lower limbs. Pharmacological interventions are not able to modify ataxia gait pattern, therefore, new approaches to rehabilitate must be studied. Treadmill locomotor training (TLT) and cerebellar transcranial direct current stimulation (ctDCS) are physical therapy techniques able to module cerebellar afferences and modify positively ataxia gait pattern. However, there is no study involving the association of these two techniques. The purpose of this study is to evaluate the effects of ctDCS associated to TLT on functional mobility in subjects with cerebellar ataxia. A randomized, sham controlled, double blind clinical trial will be performed. The subjects will be randomly allocated into two groups: (i) ctDCS associated with TLT; (ii) ctDCS sham associated with TLT. The TLT will be performed with a speed and step length progression protocol for 25 minutes. The anodal ctDCS (2 mA, 25 minutes) or sham (2mA, 30 seconds) will be applied during TLT. The functional mobility will be the primary outcome and will be evaluated through timed up and go test (TUG). Ataxia' severity, balance and fall risky, will be the secondary outcomes and will be evaluated by the scale for the assessment and rating of ataxia (SARA), balance evaluation system test (miniBest) and TUG, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Cerebellar ataxia
* Ages: 18 to 65 years;
* Gender: Both;
* Score ≥ 3 and < 8 in subscore of gait in the Scale for the Assessment and Rating of Ataxia

Exclusion Criteria:

* Individuals with other neurological disorders, postural hypotension, vestibular, visual, cardiovascular or musculoskeletal disorders that affect the performance of the proposed tests;
* Pacemaker;
* History of seizures;
* Metallic implants in the head or neck;
* Medication change during the period of study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Functional mobility | Change from baseline (T0) at 7 (T7) and 14 days (T14) after the first intervention's day
  The evaluation of the functional mobility of individuals will be performed by the Timed Up and Go test. It will analyze the time spent by the individual to get up from a chair with arms, walk for three meters and return to the chair. Longer times to performe the Timed Up and Go test mean worse functional mobility.

SECONDARY OUTCOMES:
Change in Fall risk | Change from baseline (T0) at 7 (T7) and 14 days (T14) after the first intervention's day.
  The evaluation of the functional mobility of individuals will be performed by the Timed Up and Go test. It will analyze the time spent by the individual to get up from a chair with arms, walk for three meters and return to the chair. Longer time values and step numbers represent a greater risk of falls. Time greater than 10 seconds in the test means greater risk of falling.
Change in Ataxia severity | Change from baseline (T0) at 7 (T7) and 14 days (T14) after the first intervention's day.
  The ataxia' severity will be assessed by the Scale for the Assessment and Rating of Ataxia (SARA). It consists of eight items (gait, stance, sitting, speech disturbance, finger chase, nose-finger test, fast alternating, hand movements, and heel-shin slide), where ranges from 0 to 40. Higher score mean more severe ataxia.
Change in Balance | Change from baseline (T0) at 7 (T7) and 14 days (T14) after the first intervention's day.
  The balance of individuals will be assessed through the Balance Evaluation System Test (BESt), which comprises 14 items with a score of 0-2 each from 0 (worst) to 2 (best performance), used to assess dysfunction in balance and independence in life activities daily.
Change in Patient global impression | Change from baseline (T0) at 7 (T7) and 14 days (T14) after the first intervention's day
  The patient's global impression is a questionnaire which the patient has to answer how the treatment changed his life daily activities. Patient will choose the best option that reflects their improvement in quality of life, from "no change" to "much better with differences that have made all the difference".
Adverse effects of ctDCS | 25 minutes after the beginning of stimulation
  Brunoni's questionnaire will be used to ask the patient about some possible adverse effects related to stimulations. The patient will be asked always at the end of each stimulation (real or sham).

CONTACTS AND LOCATIONS:
Locations (1):
- Kátia Monte-Silva, Recife, Pernambuco, Brazil